CLINICAL TRIAL: NCT07253272
Title: An Open-label Positron Emission Tomography (PET) Study to Demonstrate Safety, Tolerability, Receptor Occupancy, and Pharmacokinetics After a Single Oral Dose Administration of ENX-104 in Healthy Volunteers
Brief Title: A PET Study of ENX-104 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Engrail Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ENX-104-002
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENX-104 (Experimental)
  Interventions: Drug: ENX-104

INTERVENTIONS:
Drug: ENX-104 — Oral solution

SUMMARY:
The study is designed to evaluate the D2/D3 receptor occupancy (RO), safety, tolerability, and pharmacokinetics (PK) of ENX-104 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female participants (defined as assigned female at birth)

  1. Of non-childbearing potential, defined as either permanently sterilized or postmenopausal and with a negative pregnancy test
  2. Not currently breastfeeding or lactating, and not intending to initiate breastfeeding during the course of study conduct
* Biologically male participants (defined as assigned male at birth), if fertile must be willing to use a condom or remain abstinent. Participants assigned male at birth should use a highly effective method of birth control and refrain from sexual activity with partners of childbearing potential who do not use a highly effective method of birth control during the study. Participants assigned male at birth who are not surgically sterilized for at least 90 days prior to Screening and are sexually active with partner(s) of childbearing potential, must agree to refrain from sperm donation.

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the study or, in the opinion of the Investigator or Sponsor, should not participate in the study.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAE) | From Day 1 up to Day 9

CONTACTS AND LOCATIONS:
Overall Officials: David George Steel, MBChB, Principal Investigator — Parexel
Locations (1):
- Parexel London EPCU, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No